CLINICAL TRIAL: NCT07298785
Title: Peer-led Dynamic Choice HIV Prevention for Women: The Peer-led DCP Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Infectious Diseases Research Collaboration, Uganda (Other); University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25-43821; R01MH137799 (NIH)
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: HIV/AIDS
Keywords: Biomedical HIV Prevention; Peer Mentor Intervention; Uganda; Dynamic Choice HIV Prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Single-arm pilot trial to refine and pilot test the Peer-led DCP intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer-led Dynamic Choice HIV Prevention (DCP) intervention (Experimental)
  Interventions: Other: Peer-led Dynamic Choice HIV Prevention (DCP) intervention

INTERVENTIONS:
Other: Peer-led Dynamic Choice HIV Prevention (DCP) intervention — The intervention consists of peer mentor training on patient-centered choice counseling and Peer-led DCP services, and will be delivered by the peer mentor with clinician support:
  1. HIV prevention product choice with option to switch over time
  2. Rapid access to PEP from peer mentor for unplanned exposures
  3. Integration of STI testing and treatment
  4. Travel kit
  5. Phone/SMS contact for peer support

SUMMARY:
This study will refine and pilot test the Peer-led Dynamic Choice HIV Prevention (DCP) intervention in a single-arm pilot trial. The study will test the hypothesis that the Peer-led Dynamic Choice HIV Prevention intervention will be feasible and increase biomedical HIV prevention coverage in the 6 months after receipt of the Peer-led DCP intervention compared to the standard of care in the 6 months prior to intervention implementation.

DETAILED DESCRIPTION:
The overall goal of this study is to refine and pilot test a Peer-led Dynamic Choice HIV Prevention intervention tailored to women at elevated HIV risk in southwestern Uganda. We will conduct a single-arm pilot trial of the intervention enrolling approximately 60 women to assess the feasibility, acceptability, and preliminary effectiveness of the Peer-led Dynamic Choice Prevention intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years or mature or mature minor >=15 years;
2. Female sex at birth;
3. HIV negative by country-standard testing algorithm
4. Elevated risk of HIV exposure, defined as at least 1 of the following: a) eligible for PrEP based on Uganda Ministry of Health Guidelines; b) exchange of sex for goods or money in last 6 months; or c) work in bar or guesthouse

Exclusion Criteria:

* Contraindication to country-recommended PrEP regimen per national guidelines
* Participation in another HIV prevention study

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female sex at birth
Enrollment: 60 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Biomedical HIV prevention coverage | 24 weeks
  Percentage of follow-up months that a participant uses a biomedical HIV prevention product

SECONDARY OUTCOMES:
At-risk biomedical HIV prevention coverage | 24 weeks
  Percentage of at-risk follow-up months that a participant uses a biomedical HIV prevention product
Feasibility of delivery of the Peer-Led DCP intervention by peers | 24 weeks
  Proportion of participants with Peer-led DCP intervention services delivered by peer mentor

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Koss, MD, Principal Investigator — University of California, San Francisco; Jane Kabami, MPH, PhD(c), Principal Investigator — Infectious Diseases Research Collaboration
Locations (1):
- Infectious Diseases Research Collaboration, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No